CLINICAL TRIAL: NCT05231525
Title: Recovery Evaluation of Two Neuromuscular Blockade Monitoring Devices on Abductor Pollicis Muscle, the TOFScan and the Wireless WiTOF
Brief Title: Comparison of the TOFScan and the WiTOF During Recovery of Neuromuscular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WiTOF
Record Dates: First submitted 2022-01-05; First posted 2022-02-09 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Neuromuscular Residual Curarization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WiTOF (Experimental)
  Interventions: Device: WiTOF
- TOFscan (Active Comparator)
  Interventions: Device: TOFscan

INTERVENTIONS:
Device: WiTOF — Data collection on the WiTOF monitor
  Arms: WiTOF
Device: TOFscan — Data collection on the TOFscan monitor
  Arms: TOFscan

SUMMARY:
The purpose of this study is to compare two neuromuscular blockade monitors on recovery from an ATRACURIUM intra veinous injection for surgery. The TOFscan, a wired connected monitors and the WiTOF, a wireless connected monitor.

DETAILED DESCRIPTION:
The secondary objective will be to compare the performance of the two monitors on the abductor pollicis muscle with all the curarisation parameters (TOF, PTC, T4/T1R) and to assess interference occuring during the surgery which could limit the usage of a wireless monitor.

ELIGIBILITY:
Inclusion Criteria:

* All programmed surgery with intraveinous injection of ATRACURIUM
* American society of anesthesiology patient score of I, II or III
* Patient being free of tutorship or curatorship
* Acceptance of the patient after clear and loyal information

Exclusion Criteria:

* Surgery without access simultaneously to the two arms
* Emergency surgery
* Rapid sequence induction
* Usage of an other curare than ATRACURIUM
* Contraindication on ATRACURIUM usage
* Patient with pace maker
* Patient with Arné score > or = to 11
* Patient without social security coverage
* Pregnant of breastfeeding women
* Patient under social protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the neuromuscular blockade recovery after intraveinous injection of atracurium with 2 differents monitors. | During the whole period of the surgical operation maximum 8 hours
  Comparison on the obtention delay for the T4/T1 ratio superior ou equal to 90% beetween the WiTOF and the TOFScan

SECONDARY OUTCOMES:
Evaluate the performance of the monitors for the follow up of neuromuscular recovery | During the whole period of the surgical operation maximum 8 hours
  Comparison of neuromuscular blockade parameters obtained with the WiTOF and the TOFScan (TOF, PTC, T4/1R)
Number and duration of perturbation from the surgical environnement that could limit the usage of a wireless monitor | During the whole period of the surgical operation maximum 8 hours
  Assess what could perturbate the data collection on the wireless monitor

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu BOISSON, Principal Investigator — CHU de Poitiers FRANCE
Locations (1):
- CHU de Poitiers, Poitiers, France